CLINICAL TRIAL: NCT05828056
Title: Prediction on the Recurrence of Manic and Depressive Episodes in Bipolar Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002006RINA
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder; Depressive Disorder
Keywords: biomarker; Bipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BP: 100 patients with mood disorders from the psychiatric ward and outpatient services of the Department of Psychiatry, National Taiwan University Hospital
  Interventions: Device: Wearable activity tracker

INTERVENTIONS:
Device: Wearable activity tracker — Garmin smartwatch will record features, such as activities, heart rate, sleep, through smartphone App

SUMMARY:
Mood disorders (including bipolar disorder and major depressive disorder) are chronic mental disorders with high recurrent rate. The more the number of recurrence is, the worse long-term prognosis is. This study aims to establish a prediction model of recurrence of manic and depressive episodes in mood disorders, with a hope to detect recurrence relapse as early as possible for timely clinical intervention. We will adopt wearable smart watch to collect heart rate, sleep pattern, activity level, as well as emotional status for one year long in 100 patients with bipolar disorder, and annotated their mood status (i.e., manic episode, depressive episode, and euthymic state). We expect to establish prediction models to predict the recurrence of mood episodes.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 Bipolar disorder or depressive disorder
* 20~60 years old
* Willing to carry smartwatch and smartphone most of the time

Exclusion Criteria:

* Comorbid with substance use disorder
* Unable to use smartwatch and smartphone

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will recruit 100 patients with mood disorders from the psychiatric ward and outpatient services of the Department of Psychiatry, National Taiwan University Hospital. All the participants will be followed for one year to collect the daily activity level, sleep patterns, heart rate through actigraphy, as well as location, mood report, drug compliance and face photo through smartphone app that will be developed by Co-PI Lai.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and verification of mood episode prediction algorithm | 1 year
  Collected data will apply to learning algorithm, random forest, which constructs a multitude of decision trees at training time and outputting a class that is the mode of the classes of the individual trees. Performance of the trained prediction model was evaluated by assessing the model's accuracy, sensitivity, specificity, and the area under the curve. In a machine learning evaluation process, a part of data is used for model training, and the other portion is used for model testing.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
All the data in this study will be appropriately maintained with protection of privacy and confidentiality. Any personal identifiable data will be replaced by research ID number.